CLINICAL TRIAL: NCT01645384
Title: An Open-label, Randomized, Single Oral Dose, Two Way Crossover Bioequivalence Study of Atorvastatin Ca 40 mg Tablets of Dr.Reddy's With Lipitor® 40 mg Tablets of Pfizer in 74 Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Atorvastatin Calcium Tablets, 40 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01621/09-10
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Atorvastatin calcium; crossover
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin Calcium Tablets, 40 mg (Experimental): Atorvastatin Calcium Tablets, 40 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Atorvastatin Calcium Tablets, 40 mg
- Lipitor® 40 mg Tablets (Active Comparator): Lipitor® 40 mg Tablets of Pfizer Ireland Pharmaceuticals
  Interventions: Drug: Atorvastatin Calcium Tablets, 40 mg

INTERVENTIONS:
Drug: Atorvastatin Calcium Tablets, 40 mg — Atorvastatin Calcium Tablets, 40 mg of Dr. Reddy's Laboratories Limited
  Other Names: Lipitor® 40 mg Tablets

SUMMARY:
The purpose of this study is to monitor clinical status, adverse events and laboratory investigations and assess relative safety and tolerance of Atorvastatin formulations under fasting conditions.

DETAILED DESCRIPTION:
An open-label, randomized, single oral dose, two way crossover bioequivalence study to compare Atorvastatin Calcium 40 mg Tablets of Dr.Reddy's with Lipitor® 40 mg Tablets of Pfizer in 74 healthy, adult, human study participants under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* He/She should provide written informed consent.
* He/She must be a healthy adult within 18-45 years of age (inclusive).
* He/She should have a Body mass index of ≥ 18.5 kg/m2 and ≤ 25 kg/m2, with body weight not less than 50 kg.
* He/She should have a systolic blood pressure with upper limit of less than 140 mmHg and lower limit of more than or equal to 90 mm Hg. Similarly diastolic blood pressure with upper limit less than 90 mm Hg and lower limit more than or equal to 60 mmHg.
* He/She must be of normal health as determined by medical history and physical examination performed within 21 days prior to the dosing of period 1.
* He/She should have a normal ECG, chest X-ray and vital signs.
* Availability of a study volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* If study volunteer is a female and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence. or is postmenopausal for at least 1 year. or is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the study volunteers)

Exclusion Criteria:

* He/She is incapable of understanding the informed consent.
* He/She has a history of hypersensitivity or idiosyncratic reaction to study drug or any other related drug.
* He/She has any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function. Study volunteers with a history of tuberculosis, epilepsy,asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for the study.
* He/She smokes regularly more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
* He/She has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past 30 days prior to dosing in first period.
* He/She has a history of any psychiatric illness, which may impair the ability to provide written, informed consent.
* He/She has a history of alcohol or substance abuse within the last 5 years.
* He/She has clinically significant abnormal values of laboratory parameters.
* He/She has participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* He/She is unable to or likely to be non-compliant with protocol requirements or restrictions.
* He/She, in whom study drug is contraindicated for medical reasons
* He/She is intolerant to venipuncture.
* Female volunteer who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing.
* Female volunteer demonstrates a positive pregnancy screen. Each female study volunteer will be screened for pregnancy at screening, check-in each study period. Study volunteer with a positive or inconclusive result will be withdrawn from the study.
* Female volunteer is currently breast feeding. Female study volunteer who is pregnant, breast-feeding or who is likely to become pregnant during the study will not be allowed to participate. Female study volunteer of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or she will not be allowed to participate.
* He/She has a positive urine screen for drugs of abuse at the time of admission check-in for each period will be excluded from the study.
* He/She, who meets the inclusion and exclusion criteria, will be verified by medical investigator as per source documents duly authenticated by them reflecting clinical judgment as and when required

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose at 0.00, 0.167, 0.333, 0.50, 0.667, 0.833, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 2.75, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 hours and 48.00 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sudarshan Vishwanath, MD, Principal Investigator — Vimta Labs Limited
Locations (1):
- Vimta Labs Limited, Hyderabad, Andhra Pradesh, India